CLINICAL TRIAL: NCT07086911
Title: The Impact of Tosylate Remimazolam on Oxygenation and Postoperative Cognitive Function in Elderly Patients Undergoing Thoracoscopic Lobectomy
Brief Title: The Impact of Remimazolam Tosilate on Oxygenation and Postoperative Cognitive Function in Elderly Patients Undergoing Thoracoscopic Lobectomy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jinqiao Qian (Other)
Responsible Party: Sponsor-Investigator, Jinqiao Qian, deputy director, First Affiliated Hospital of Kunming Medical University
Organization: First Affiliated Hospital of Kunming Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZKL-KY20241015-78
Record Dates: First submitted 2025-06-27; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Remimazolam Besylate; Thoracoscopic Lobectomy; Oxygenation; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — remimazolam; Propofol

STUDY DESIGN:
Intervention Model Description: Remimazolam group (Group R): After intubation, remimazolam was maintained at a pump rate of 1-2mg/kg/h until 10 minutes before the end of the surgery. Propofol group (Group P): After intubation, propofol was maintained at a pump rate of 4-10mg/kg/h until 10 minutes before the end of the surgery.
  Remimazolam combined with propofol group (Group C): After intubation, it was maintained at 0.3-1mg/kg/h of remimazolam +3-6 mg/kg/h of propofol until 10 minutes before the end of the operation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person responsible for grouping; Data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam Group (Group R) (Experimental): After intubation, remimazolam was maintained at a pump rate of 1-2mg/kg/h until 10 minutes before the end of the operation.
  Interventions: Drug: Remimazolam
- Propofol group (Group P) (Active Comparator): After intubation, propofol was maintained at a pump rate of 4-10mg/kg/h until 10 minutes before the end of the operation
  Interventions: Drug: Propofol
- Remimazolam combined with propofol group (Group C) (Experimental): After intubation, remimazolam at a dose of 0.3-1mg/kg/h and propofol at a dose of 3-6 mg/kg/h were maintained until 10 minutes before the end of the operation
  Interventions: Drug: Remimazolam; Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam group (Group R) : After intubation, remimazolam was maintained at a pump rate of 1-2mg/kg/h until ten minutes before the end of the operation.
  Group C (remimazolam combined with propofol): After intubation, maintain with 0.3-1 mg/kg/h of remimazolam and 3-6 mg/kg/h of propofol until 10 minutes before the end of surgery.
  Arms: Remimazolam Group (Group R); Remimazolam combined with propofol group (Group C)
Drug: Propofol — Propofol group (Group P) : After intubation, propofol was maintained at a pump rate of 4-10mg/kg/h until surgery ten minutes before the end.
  Group C (remimazolam combined with propofol): After intubation, maintain with 0.3-1 mg/kg/h of remimazolam and 3-6 mg/kg/h of propofol until 10 minutes before the end of surgery.
  Arms: Propofol group (Group P); Remimazolam combined with propofol group (Group C)

SUMMARY:
Background: During thoracoscopic lobectomy in elderly patients, one-lung ventilation (OLV) is a common procedure. However, this process is prone to cause hypoxemia and postoperative cognitive dysfunction (POCD), which seriously affect the postoperative recovery and prognosis of patients. At present, there is still a need for further exploration and optimization of effective anesthetic drugs and regimens to improve intraoperative oxygenation and reduce the occurrence of POCD in such patients. Remimazolam besylate, as a novel anesthetic drug, has not yet had its advantages in thoracoscopic surgery in elderly patients fully clarified. This study is conducted to explore its effects on oxygenation and postoperative cognitive function in this specific surgical setting, so as to provide new references for clinical drug use and improve the perioperative management and postoperative outcomes of elderly patients.

Objective:To mainly investigate the effects of remimazolam besylate on oxygenation and intrapulmonary shunting during one-lung ventilation in elderly patients undergoing thoracoscopic surgery, as well as its impact on postoperative cognitive dysfunction.

Research Content:The research content includes the observation and evaluation of oxygenation index, shunt fraction, cognitive function status, intraoperative conditions (such as OLV duration, blood loss, etc.),hemodynamic indicators, blood gas analysis indicators, serum indicators, and postoperative recovery status (such as postoperative sedation, pain, adverse reactions, pulmonary complications, hospital stay duration, etc.) in elderly patients undergoing thoracoscopic lobectomy.

Research Methods:

Study Design: A randomized controlled study will be adopted. Case Selection: Inclusion Criteria: Patients aged 65-75 years old, with a BMI of 18-30 kg/m², ASA classification of I-III, no contraindications to related drugs, and consent from the patient and their family to participate in the study and sign the informed consent form, who are scheduled for thoracoscopic surgery under general anesthesia at the First Affiliated Hospital of Kunming Medical University from December 2024 to December 2025, will be selected. Exclusion Criteria: Patients with severe arrhythmias, preoperative respiratory tract infections, central nervous system diseases, hepatic or renal insufficiency, immune system diseases, a history of preoperative radiotherapy or chemotherapy, communication barriers, etc., will be excluded. Exclusion Criteria: Patients with OLV duration less than 60 minutes or conversion to thoracotomy, intraoperative blood loss greater than 1000 ml, and those transferred to the ICU after surgery will be excluded.

Grouping and Anesthesia Methods: Patients will be randomly divided into three groups: Remimazolam Group (R Group), Propofol Group (P Group), and Remimazolam Combined with Propofol Group (C Group), with 50 cases in each group. After anesthesia induction, the three groups will be maintained with different drugs and doses until 10 minutes before the end of the surgery, while remifentanil will be combined, and the infusion rate of the drugs will be adjusted according to the BIS value.

Data Collection: Detailed records will be kept of the patient's general information, intraoperative conditions, perioperative cardiovascular reactions, blood gas analysis indicators, serum indicators, as well as postoperative cognitive function assessment, sedation and pain assessment, adverse reactions, and complications.

Sample Size Calculation: Based on the oxygenation index at 60 minutes of OLV, which is the primary endpoint, and in combination with relevant literature and statistical requirements, the sample size for each group is calculated to be 58. Considering the dropout and withdrawal rates, the final sample size for each group is determined to be 70.

Statistical Analysis: SPSS 27.0 software will be used. Normal distribution measurement data, non-normal distribution measurement data, and count data will be analyzed using independent sample t-test, Wilcoxon rank-sum test, and chi-square test or Fisher's exact probability method, respectively. A P value less than 0.05 will be considered statistically significant.

Technical and Feasibility Assurance: Relying on the clinical resources and technical platform of the First Affiliated Hospital of Kunming Medical University, as well as the research team's proficiency in thoracic anesthesia techniques and the operation of related equipment, the smooth conduct of the study will be ensured.

DETAILED DESCRIPTION:
This study aims to investigate the effects of remimazolam besylate on oxygenation and postoperative cognitive function in elderly patients undergoing thoracoscopic lobectomy with one-lung ventilation. This randomized controlled study selected 150 elderly patients aged 65 to 75 years, with a BMI of 18 to 30 kg/m², ASA classification of I to III, no contraindications to related drugs, and informed consent, who were scheduled for thoracoscopic surgery under general anesthesia at the First Affiliated Hospital of Kunming Medical University from December 2024 to December 2025. Patients with severe arrhythmias, preoperative respiratory tract infections, central nervous system diseases, etc., were excluded. Patients were randomly divided into three groups: Remimazolam Group (R Group), Propofol Group (P Group), and Remimazolam Combined with Propofol Group (C Group), with 50 cases in each group. After anesthesia induction, the three groups were maintained with different drugs and doses until 10 minutes before the end of the surgery, while remifentanil was combined, and the infusion rate of the drugs was adjusted according to the BIS value. The observed indicators included oxygenation index, shunt fraction, cognitive function status, intraoperative conditions, hemodynamic indicators, blood gas analysis indicators, serum indicators, and postoperative recovery status, etc. The study results showed that the remimazolam group had certain advantages in intraoperative oxygenation, a relatively lower incidence of postoperative cognitive dysfunction, and no significant increase in postoperative adverse reactions. The results of this study indicate that remimazolam besylate has certain application advantages in thoracoscopic surgery in elderly patients, can improve intraoperative oxygenation, reduce the risk of postoperative cognitive dysfunction, and provide a new reference for the selection of clinical anesthetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoscopic surgery under general anesthesia at the First Affiliated Hospital of Kunming Medical University;
* Age 65 to 75 years old;
* BMI18-30 kg/m ²;
* ASA grades I to III;
* There are no contraindications to any related drugs;
* Both the patient and their family members agreed to participate in this study and signed the informed consent form

Exclusion Criteria:

* Patients with severe sinus bradycardia (heart rate <50 beats per minute) and atrioventricular block;
* Respiratory tract infection and the use of non-steroidal anti-inflammatory drugs or hormone drugs within 2 weeks before the operation;
* Those with central nervous system and psychological disorders;
* Have taken anticholinergic drugs, anticonvulsants, anti-anxiety drugs, antidepressants, etc. in the past half year;
* Severe liver and kidney dysfunction and immune system diseases, uncontrolled hypertension and diabetes;
* History of preoperative radiotherapy and chemotherapy;
* Patients with communication barriers who are unable to cooperate to complete the test;
* The OLV < 60 min or interim thoracotomy patients;
* Intraoperative blood loss > 1500ml;
* Patients transferred to the ICU ward after the operation.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
(1)The oxygenation index and shunt fraction of the patients at different times; | perioperative
  (1) Oxygenation index and shunt fraction of patients at different times: before one-lung ventilation (T1), 30 minutes of one-lung ventilation (T2), 60 minutes of one-lung ventilation (T3).
(2)Cognitive function situation | within 7days following surgery
  (2) cognitive function: POCD occurs within 7 days following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jinqiao Qian, doctor, Study Director — First Affiliated Hospital of Kunming Medical University
Locations (1):
- The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
Patient Basic Information: Age, gender, ASA classification, BMI, surgical approach, operative side, preoperative baseline pulmonary function, etc.
  Intraoperative Conditions: Duration of one-lung ventilation (OLV), blood loss, volume of fluid infusion, remimazolam dosage, propofol dosage, remifentanil dosage, urine output, ephedrine dosage, atropine dosage, incidence of hypoxemia, etc.
  Perioperative Cardiovascular Response: Heart rate (HR), mean arterial pressure (MAP), pulse oxygen saturation (SpO₂) recorded at the following time points: upon entering the operating room (T0), before OLV initiation (T1), 30 minutes after OLV initiation (T2), 60 minutes after OLV initiation (T3), before extubation (T4), and 5 minutes after extubation (T5).
  Blood Gas Analysis Indicators:Arterial and central venous blood gas analyses were performed on all patients at T1 (before OLV), T2 (30 min after OLV), and T3 (60 min after OLV). Recorded parameters included: airway plateau pressure (Pplat)and so on.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The sharing period is from August 2025 to August 2026.
Access Criteria: All researchers have access to the IPD and supporting information. They can access the study protocol design, as well as subsequent data collection and analysis results. They can search for this information on this website by entering the study title.

DOCUMENTS (2):
  • Study Protocol (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT07086911/Prot_000.pdf
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT07086911/ICF_001.pdf